CLINICAL TRIAL: NCT04800653
Title: The Effect of Stellate Ganglion Block on Postoperative Sleep Disturbance and Cognitive Function in Elderly Surgical Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yangzhou University (Other)
Responsible Party: Principal Investigator, Zhuan Zhang, Director, Yangzhou University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 202103101
Record Dates: First submitted 2021-03-11; First posted 2021-03-16 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Stellate Ganglion Block
Keywords: Delirium; Cognitive Dysfunction; Sleep Disorders
MeSH Terms: conditions — Delirium; Cognitive Dysfunction; Sleep Wake Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stellate ganglion block (Experimental): Before the operation, the left stellate ganglion block was performed, and 0.375% ropivacaine 5ml was injected into the stellate ganglion.
  Interventions: Procedure: Stellate ganglion block
- Control (No Intervention): Do nothing

INTERVENTIONS:
Procedure: Stellate ganglion block — Find the position of the stellate ganglion under ultrasound guidance, and inject 0.375% ropivacaine near the stellate ganglion to block the sympathetic nerves in the upper chest and head and neck
  Arms: Stellate ganglion block

SUMMARY:
Postoperative delirium is an acute state of confusion, which is characterized by changes in attention and cognitive functions and fluctuations in consciousness; postoperative cognitive dysfunction is a common central nervous system complication in elderly patients after surgery, often manifested as memory, Obstacles in abstract thinking and orientation are accompanied by a decline in social activity ability. Postoperative delirium and cognitive dysfunction can prolong hospital stay, increase medical expenses, affect postoperative functional recovery, and even increase postoperative mortality. Sleep disorders are a group of diseases that affect the ability to sleep well regularly and cause severe impairment of social and occupational functions. Stellate ganglion block is a selective sympathetic ganglion block, in which a local anesthetic is injected into the loose connective tissue of the neck including the stellate ganglion. There are complex connections between stellate ganglia and multiple brain regions in the brain, which can improve postoperative delirium, cognitive function and sleep disturbance to a certain extent, and have certain guiding significance for postoperative rehabilitation of elderly patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 60 years;
2. ASA grade I-III;
3. Operative time ≥ 2 h for laparoscopic radical resection of a suspected; gastrointestinal malignancy.

Exclusion criteria :

1. Patient's lack of consent to participate;
2. Known allergy to anesthetic drugs;
3. History of psychiatric or neurological disease(s);
4. Long-term use of opioids or sedative-hypnotic drugs;
5. Previous or planned neurosurgical procedures;
6. contraindications to epidural anesthesia;
7. Hearing or visual impairment that precludes scale assessment.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-07-12 (Actual)

PRIMARY OUTCOMES:
Changes in the level of Mini-Men-tal State Examination scale score | The day before surgery and 1,2,3,5,7 days after surgery
  Assess the cognitive function of the patient by asking questions on the patient scale
Changes in the level of actigraphy | The 1st night before the operation and the 1st, 2nd and 3rd nights postoperatively
  Through the actigraphy, monitor the patient's sleep quality
Changes in the level of Pittsburgh sleep quality index | The day before surgery and 1,2,3,5,7 days
  Assess the patient's sleep quality by asking questions on the scale

SECONDARY OUTCOMES:
Changes in the level of IL-1 | Preoperative, 6 am on the first day after surgery, 6 am on the third day after surgery
  The outcome above should be measured at the time Preoperative, 6 am on the first day after surgery, 6 am on the third day after surgery
Changes in the level of Systolic Blood Pressure/Diastolic Blood Pressure(Mean Arterial Pressure) | Baseline (Before induction), immediately before intubation, immediately after intubation, at the beginning of the operation, 1 hour after the beginning of the operation, and immediately after extubation at the end of the operation
  The outcome above should be measured at the time Before induction, immediately before intubation, immediately after intubation, at the beginning of the operation, 1 hour after the beginning of the operation, and immediately after extubation at the end of the operation
Local cerebral Oxygen Saturation | Collected every 15 minutes before induction of anesthesia to 1 hour after the end of anesthesia
  The outcome above should be measured Local cerebral oxygen saturation meter
Changes in the level of IL-10 | Preoperative, 6 am on the first day after surgery, 6 am on the third day after surgery
  The outcome above should be measured at the time Preoperative, 6 am on the first day after surgery, 6 am on the third day after surgery
Changes in the level of IL-6 | Preoperative, 6 am on the first day after surgery, 6 am on the third day after surgery
  The outcome above should be measured at the time Preoperative, 6 am on the first day after surgery, 6 am on the third day after surgery
Changes in the level of Melatonin | Preoperative, 6 am on the first day after surgery, 6 am on the third day after surgery
  The outcome above should be measured at the time Preoperative, 6 am on the first day after surgery, 6 am on the third day after surgery
Changes in the level of Heart Rate | Baseline (Before induction), immediately before intubation, immediately after intubation, at the beginning of the operation, 1 hour after the beginning of the operation, and immediately after extubation at the end of the operation
  The outcome above should be measured at the time Before induction, immediately before intubation, immediately after intubation, at the beginning of the operation, 1 hour after the beginning of the operation, and immediately after extubation at the end of the operation
Changes in the level of Oxygen saturation | Baseline (Before induction), immediately before intubation, immediately after intubation, at the beginning of the operation, 1 hour after the beginning of the operation, and immediately after extubation at the end of the operation
  The outcome above should be measured at the time Before induction, immediately before intubation, immediately after intubation, at the beginning of the operation, 1 hour after the beginning of the operation, and immediately after extubation at the end of the operation
Changes in the value and waveform of Narcotrend | Baseline (Before induction), immediately before intubation, immediately after intubation, at the beginning of the operation, 1 hour after the beginning of the operation, and immediately after extubation at the end of the operation
  The outcome above should be measured at the time Before induction, immediately before intubation, immediately after intubation, at the beginning of the operation, 1 hour after the beginning of the operation, and immediately after extubation at the end of the operation
Changes in the level of S100-β | Preoperative, 6 am on the first day after surgery, 6 am on the third day after surgery
  The outcome above should be measured at the time Preoperative, 6 am on the first day after surgery, 6 am on the third day after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- the Affiliated Hospital of Yangzhou University, Yangzhou, Jiangsu, China

REFERENCES:
- [Derived] Yan S, Wang Y, Yu L, Xia W, Xue F, Yu Y, Yuan B, Li N, Li H, Liang H, Ma J, Zhang Z. Stellate ganglion block alleviates postoperative sleep disturbance in patients undergoing radical surgery for gastrointestinal malignancies. J Clin Sleep Med. 2023 Sep 1;19(9):1633-1642. doi: 10.5664/jcsm.10632. PMID 37128727